CLINICAL TRIAL: NCT06189664
Title: Evaluation of the Effectiveness of Intraoperative Frozen Section on the Treatment of Suspected Gallbladder Cancer
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: Gen_17/2020
Record Dates: First submitted 2023-12-19; First posted 2024-01-03 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Gallbladder Cancer
MeSH Terms: conditions — Gallbladder Neoplasms | interventions — Frozen Sections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Frozen section — Frozen section analysis

SUMMARY:
Evaluate the effectiveness of intra-operative frozen section in the treatment of gallbladder cancer.

The study will be looking in to identify if intraoperative frozen section is a viable method to intraoperatively evaluate the presence of adenocarcinoma and the depth of its invasion and if the information given by frozen section is enough to modify the operative strategy.

ELIGIBILITY:
Inclusion Criteria:

- Patients with suspected GB cancer

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with suspected GB Cancer
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Detection of adenocarcinoma | immediately during frozen section

REFERENCES:
- [Derived] Banh S, Fehervari M, Flod S, Soleimani-Nouri P, Leyte Golpe A, Ahmad R, Pai M, Spalding DRC. Single stage management of suspected gallbladder cancer guided by intraoperative frozen section analysis: a retrospective cohort study. Int J Surg. 2024 Oct 1;110(10):6314-6320. doi: 10.1097/JS9.0000000000001456. PMID 38704628